CLINICAL TRIAL: NCT04672174
Title: Cognitive Screening of Patients with Hearing Loss
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UniversitätsSpital Zürich
Record Dates: First submitted 2020-11-19; First posted 2020-12-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of hearing loss on dementia (Other): Effect of hearing loss on dementia, collected with a standardized questionnaire
  Interventions: Diagnostic Test: Questionnaire: DemTect

INTERVENTIONS:
Diagnostic Test: Questionnaire: DemTect — Questionnaire is handed out to subjects

SUMMARY:
Hearing loss and cognitive impairment both appear in elderly patients. The goal was to use a modified screening method added to already established cognitive tests to obtain a standardized test for detection of cognitive impairment in patients with hearing loss.

The aim of this study is to collect data with neuropsychological tests using questionnaires and to determine cognitive impairment in patients with hearing loss.

The collected data will be evaluated using SPSS 23. The corrected item-total correlation and item difficulty of the item DemTectEar will be assessed by item analysis / Cronbachs' Alpha. For further evaluation and comparisons two-sided t-tests with a level of significance 0.05 or Mann-Whitney-U-tests will be performed.

DETAILED DESCRIPTION:
Cognitive impairment and dementia are a growing health-care problem in our society. The prevalence of dementia is still estimated to grow drastically and reach over a 100 million world-wide by the year 2050. To address this problem there are numerous neuropsychological screening methods, for example the mini-mental state examination (MMSE) or the DemTect.

Another age-dependent problem is the increasing hearing impairment. Furthermore, studies have shown that hearing loss is associated with cognitive decline and may accelerate the process. Nevertheless, there is no specific cognitive screening method for patients with a sensory hearing loss.

This study aims to obtain a specifically modified version of the general DemTect called DemTectEar for patients with pre-existing hearing loss. Such a screening method would lead to earlier detection, earlier therapy and thereby to deceleration of cognitive decline.

Patient charts are screened to identify possible participants. They are contacted to participate in the study during regular clinical follow-up consultations or are contacted by phone or mail.

The investigators will explain to each participant the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits and any discomfort it may entail. Each participant will be informed that the participation in the study is voluntary and that he or she may withdraw from the study at any time and that withdrawal of consent will not affect his or her subsequent medical assistance and treatment.

The participant will be informed that his or her medical records may be examined by authorised individuals other than their treating physician.

All participants for the study will be provided a participant information sheet and a consent form describing the study and providing sufficient information for participant to make an informed decision about their participation in the study. Enough time, a few days or more if required, will be given to the participant to decide whether to participate or not.

The formal consent of a participant, using the approved consent form, will be obtained before the participant is submitted to any study procedure.

The consent form will be signed and dated by the investigator or his designee at the same time as the participant sign. A copy of the signed informed consent will be given to the study participant. The consent form will be retained as part of the study records.

Study procedures

The overall duration of the study is planned to be 12 months starting with the recruitment period on September 2019. The study duration for each patient is planned to be approximately 60 min, in which each patient will be undergoing a series of neuropsychological tests and questionnaires such as:

DemTectEar Mini Mental State Examination (MMSE) F-A-S Becks Depressions-Inventar (BOI-V) Bayer-Activities of Daily Living Scale-Skala (B-ADL Skala) Trail Making Test (TMT) Rey-Osterrieth Complex Figure Test - Copy and Recall (ROCFT) Mini-q Test Nürnberger-Alters-Inventar Test (NAI-Labyrinth) Subtest 4 of the Leistungsprüfsystem für 50+ (LPS50+) Subtest 6 of the Leistungsprüfsystem für 50+ Verbaler Lern- und Merkfähigkeitstest (VLMT) Geriatrische Depressionsskala (GDS)

Statistical analysis plan and sample size calculation The collected data will be evaluated using SPSS 23. The corrected item-total correlation and item difficulty of the item DemTectEar will be assessed by item analysis / Cronbachs' Alpha. For further evaluation and comparisons two-sided t-tests with a level of significance 0.05 or Mann-Whitney-U-tests will be performed. The primary endpoint consists of a cut-off score between age-appropriate cognitive capability and cognitive impairment.

In total, 200 control subjects, 50 patients with a hearing loss and 50 patients with visual impairment will be included for analysis. The majority of these patients is recruited in Köln, and only 20 patients with hearing impairment are investigated in Zürich.

ELIGIBILITY:
Inclusion Criteria:

* - Age 50 - 90
* Measurable hearing loss
* Sufficient knowledge of german
* Ability to consent

Exclusion Criteria:

* Age < 50 or >90
* No measurable hearing loss
* Present or past alcohol or drug abuse
* Clinically relevant depressive symptoms
* lnability to consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire to assess effect of hearing loss on memory (DemTect) | 2 years
  Effect of hearing loss on memory

CONTACTS AND LOCATIONS:
Overall Officials: Christof Roosli, Principal Investigator — UniversitätsSpital Zürich, ORL-Klinik
Locations (1):
- Andrea Kegel, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No